CLINICAL TRIAL: NCT02296905
Title: Pharmacokinetics and Safety of ABT-493 and/or ABT-530 in Subjects With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M13-604
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir; pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group I (Experimental): Subjects with mild hepatic impairment
  Interventions: Drug: ABT-493; Drug: ABT-530
- Group II (Experimental): Subjects with moderate hepatic impairment
  Interventions: Drug: ABT-493; Drug: ABT-530
- Group III (Experimental): Subjects with severe hepatic impairment
  Interventions: Drug: ABT-493; Drug: ABT-530
- Group IV (Experimental): Subjects with normal hepatic function
  Interventions: Drug: ABT-493; Drug: ABT-530

INTERVENTIONS:
Drug: ABT-493 — Up to 2 single doses of ABT-493 will be given orally in combination with ABT-530.
Drug: ABT-530 — Up to 3 single doses of ABT-530 will be given orally alone or in combination with ABT-493.

SUMMARY:
This is an open-label, single-dose study designed to assess the pharmacokinetics and safety of ABT-493 and/or ABT-530 in subjects with impaired hepatic function and compare them to those in subjects with normal hepatic function.

Twenty-four subjects will be selected and enrolled according to the subject selection criteria: 6 subjects with mild stable chronic hepatic impairment (Group I), 6 subjects with moderate stable chronic hepatic impairment (Group II), 6 subjects with severe stable chronic hepatic impairment (Group III) and 6 subjects with normal hepatic function (Group IV).

ELIGIBILITY:
Inclusion Criteria: All Subjects

* If female, subject must be either postmenopausal for at least 2 years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy).
* Females must have negative results for pregnancy test performed:

  * At Screening on a urine specimen obtained within 28 days prior to initial study drug administration, and
  * On a serum sample obtained on Study Day -1 of Period 1.
* Males must be surgically sterile or practicing at least one of the following methods of birth control (sperm donation within the study period is not allowed):

  * Abstinence
  * Partner(s) using an Intrauterine Device (IUD)
  * Partner(s) using oral, injected, or implanted methods of hormonal contraceptives
  * Subject and/or partner(s) using double-barrier method.

Subjects with Normal Hepatic Function

In addition to the inclusion criteria above for all subjects, the following criteria must be met for subjects with normal hepatic function enrolled in Group IV:

* Judged to be in general good health based upon the results of a medical history, physical examination, laboratory profile (including liver function parameters within the limits of normal) and 12-lead electrocardiogram (ECG).
* Negative hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (HCV Ab) test results.
* Body Mass Index (BMI) is ≥ 18 to < 38 kg/m2, inclusive.

Subjects with Hepatic Impairment

In addition to the inclusion criteria for all subjects, the following criteria must be met for all subjects with hepatic impairment enrolled in Groups I, II and III:

* Judged to be in stable condition and acceptable for study participation based upon the results of a medical history, physical examination, laboratory profile and ECG.
* BMI is ≥ 18 to < 38 kg/m2, inclusive, for subjects with hepatic impairment without ascites or subjects with subclinical ascites detected only by ultrasound or other imaging. For subjects with hepatic impairment and clinically significant ascites, BMI is permitted in the range between ≥ 18 to < 40 kg/m2, inclusive.
* Child-Pugh classification of Categories A (mild), B (moderate), or C (severe).
* Medical history of chronic liver disease including and not limited to chronic hepatitis B, history of alcoholic liver disease and chronic hepatitis C.
* Presence of clinically significant hepatic impairment as indicated by either:

  1. Evidence of liver cirrhosis OR
  2. Medical history of at least one of the following criteria:

     * Clinical diagnosis of liver disease
     * Total bilirubin, > 2 mg/dl, with indirect/direct ratio < 1 or prolonged prothrombin time elevation > 1.7 or an albumin value below the lower limit of the laboratory reference range and excluding non-hepatic causes of the previous laboratory abnormalities.

Exclusion Criteria: - History of significant sensitivity to any drug.

* Pregnant or breastfeeding female.
* Recent (6-month) history of drug or alcohol abuse.
* Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM) or human immunodeficiency virus antibody (HIV Ab). Negative HIV status will be confirmed at Screening and the results will be maintained confidentially by the study site.
* Detectable HCV RNA.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall measurement of pharmacokinetic parameter values of ABT-493 and ABT-530 | 7 days
  Pharmacokinetic parameter values include the maximum plasma concentration (Cmax), the terminal phase elimination rate constant (B), the area under the plasma concentration-time curve (AUC) from time 0 to time of the last measurable concentration (AUCt).
Overall measurement of safety parameters | Up to 38 days
  Measurement of safety parameters include physical examinations, clinical laboratory tests, 12-lead ECGs (electrocardiograms) and vital signs.
Number of subjects with adverse events | Up to 58 days

CONTACTS AND LOCATIONS:
Overall Officials: David Pugatch, MD, Study Director — AbbVie
Locations (4):
- United States (3):
  - Site Reference ID/Investigator# 130589, Miami, Florida
  - Site Reference ID/Investigator# 130591, Orlando, Florida
  - Site Reference ID/Investigator# 130588, San Antonio, Texas
- Site Reference ID/Investigator# 130590, Grafton, New Zealand